CLINICAL TRIAL: NCT03086590
Title: BODY COMPOSITION, PERIPHERAL MUSCULAR FORCE, KINEMATIC THORACIC-ABDOMINAL, VENTILATORY METABOLIC RESPONSE, DIAPHRAGM MOBILITY AND THICKNESS PREDICTION OF OBSTRUCTION LEVEL OF COPD?
Brief Title: EVALUATION OF RESPIRATORY MECHANICS AND FUNCTIONALITY IN PATIENTS WITH CHRONIC OBSTRUCTIVE PULMONARY DISEASE
Status: Completed | Type: Observational
Sponsor: Universidade Federal de Pernambuco (Other)
Responsible Party: Principal Investigator, Rodrigo Viana Correia de Souza, Principal Investigator, Universidade Federal de Pernambuco
Other Study IDs: UFPE-M1
Record Dates: First submitted 2017-03-09; First posted 2017-03-22 (Actual); Last update posted 2018-11-07 (Actual); Status verified 2018-11

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: Body composition; Ultrasound; Chronic Pulmonary Obstructive Disease; Respiratory muscles
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional

GROUPS / COHORTS (4):
- Group 1: COPD mild. The individuals allocated to this group have FEV1 ≥ 80% predicted.
- Group 2: COPD Moderate. The individuals allocated to this group have 50% ≤ FEV1 < 80% predicted.
- Group 3: COPD Severe. The individuals allocated to this group have 30% ≤ FEV1 < 50% predicted.
- Group 4: COPD Very severe. The individuals allocated to this group have FEV1 < 30% predicted.

SUMMARY:
To associate a lean mass, peripheral muscle strength, kinematic thoracic-abdominal, respiratory metabolic response, mobility and diaphragmatic thickness, verifying its relation with the obstruction level of COPD

DETAILED DESCRIPTION:
Individuals with COPD present restriction in their daily lives due to changes and bodily disorders promoted by the disease, such as changes in types of muscle fibers and chronic inflammatory process, causing a low level of physical activity and quality of life, besides being closely Related to the need for hospitalizations and increased mortality. A cross-sectional study with a convenience sample was performed at the Laboratory of Cardiopulmonary Physiotherapy of the Federal University of Pernambuco during the period from December 2016 to February 2018. As measurements of body composition were performed with a bio-balance scale, Evaluation of the peripheral muscle strength will be used the dynamometer, a load cell and electromyography, a kinematic thoracic-abdominal will be measured by optoelectronic plethysmography, a respiratory metabolic response will be verified during the 6-minute walk test using the gas analyzer, and for evaluation of mobility and diaphragmatic thickness are used on ultrasound associated with pneumotachograph.

ELIGIBILITY:
Inclusion Criteria:

* Young adults, adults and elderly subjects

Exclusion Criteria:

* Others respiratory diseases;
* Heart diseases;
* Those who are in some previous training program or rehabilitation;

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with Chronic Obstructive Pulmonary Disease, selected at the Hospital das Clínicas of the Federal University of Pernambuco, Hospital Otávio de Freitas and Pharmacy of the State of Pernambuco.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2016-11-01 (Actual); Primary Completion 2018-02-01 (Actual); Study Completion 2018-03-01 (Actual)

PRIMARY OUTCOMES:
Fat-free mass | Baseline
  Mass of the human body disregarding fat.
Quadriceps Force | Baseline
  Quadriceps muscle strength measured during maximum voluntary contraction.
Handgrip strength | Baseline
  Maximum voluntary manual holding force.
Total chest wall volume | Baseline
  Total volume resulting from the sum of the volume of the pulmonary compartment of the costal, abdominal gradient of the costal and abdominal beds.
Oxygen uptake | Baseline
  Consumption of oxygen during an effort.
Diaphragm mobility | Baseline
  It is the diaphragmatic movement from the end of the expiration until the end of the inspiration, being able to be realized in tidal volume or starting from the total pulmonary capacity.
Diaphragm thickness | Baseline
  Defined as a corpulence of the diaphragm muscle

CONTACTS AND LOCATIONS:
Locations (1):
- Universidade Federal de Pernambuco, Recife, Pernambuco, Brazil